CLINICAL TRIAL: NCT00082927
Title: A Multicentre Randomised Trial Of Single Dose Radiotherapy Compared To Ibandronate For Localised Metastatic Bone Pain
Brief Title: Single-Dose Local Radiation Therapy Compared With Ibandronate in Treating Patients With Localized Metastatic Bone Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CRUK-NCRI-RT-02-01; CDR0000361728 (Registry Identifier: PDQ (Physician Data Query)); EU-20224; RIB; ISRCTN86185157
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Metastatic Cancer; Pain; Prostate Cancer
Keywords: stage IV prostate cancer; bone metastases; pain; recurrent prostate cancer
MeSH Terms: conditions — Neoplasm Metastasis; Pain; Prostatic Neoplasms | interventions — Ibandronic Acid

INTERVENTIONS:
Drug: ibandronate sodium

SUMMARY:
RATIONALE: Ibandronate may be effective in reducing bone pain caused by metastatic cancer. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether ibandronate is more effective than standard treatment with radiation therapy in treating metastatic bone pain.

PURPOSE: This phase III randomized clinical trial is studying ibandronate to see how well it works compared to single-dose local radiation therapy in treating patients with localized metastatic bone pain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare pain response at 4 and 12 weeks post-treatment in patients with localized metastatic bone pain treated with single-dose ibandronate vs single-dose local radiotherapy .

Secondary

* Compare the quality of life of patients treated with these regimens.
* Correlate urinary markers of osteoclast activity (pyridinoline and deoxypyridinoline) with the clinical outcome of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, crossover, multicenter study. Patients are stratified according to primary tumor type and participating center. Patients are randomized into 1 of 2 treatment arms.

* Arm I: Patients receive a single dose of local radiotherapy to the site of pain (8Gy/1f).
* Arm II: Patients receive a single dose of ibandronate IV over 15 minutes. Patients who do not achieve a partial or complete response at 4 weeks crossover to the alternate arm.

Quality of life is assessed at baseline and then at 4 and 12 weeks. Pain is assessed at baseline, at 4, 8, and 12 weeks, and then at 6 months.

Patients are followed at 4, 8, and 12 weeks and then at 6 and 12 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 470 patients (235 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary prostate cancer OR sclerotic bone metastases (for patients with serum prostate-specific antigen > 100 ng/mL)
* Radiologically confirmed bone metastases by plain x-ray, isotope scan, CT scan, or MRI
* Clinical diagnosis of metastatic bone pain for which radiotherapy is indicated
* Single localized metastatic bone pain AND receiving optimal analgesics and adjuvant drugs, including non-steroidal anti-inflammatory drugs, unless contraindicated
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Over 18

Sex

* Male

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Creatinine ≤ 3.0 mg/dL
* No hypercalcemia (corrected calcium > 10.8 mg/dL)
* No hypocalcemia (corrected calcium < 8.2 mg/dL)

Other

* No known hypersensitivity to ibandronate or other bisphosphonates
* No history of aspirin-sensitive asthma
* Able to comply with pain chart and quality of life assessments

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior change in systemic chemotherapy
* No prior high-dose chemotherapy (dose intensity > 3 times standard dose)

Endocrine therapy

* More than 4 weeks since prior change in hormonal therapy

Radiotherapy

* See Disease Characteristics
* No prior external beam radiotherapy to index site
* No prior systemic radioisotope therapy (e.g., strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium)

Surgery

* Not specified

Other

* More than 6 months since prior bisphosphonate treatment
* More than 4 weeks since prior aminoglycoside antibiotics
* More than 30 days since prior investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2003-04; Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Purnell — Cancer Research UK; Katherine Monson — Cancer Research UK
Locations (52):
- United Kingdom (52):
  - William Harvey Hospital, Ashford-Kent, England
  - North Devon District Hospital, Barnstaple, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Royal United Hospital, Bath, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Queen's Hospital, Burton-on-Trent, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Cumberland Infirmary, Carlisle, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Mayday University Hospital, Croydon, England
  - Russells Hall Hospital, Dudley, England
  - Eastbourne District General Hospital, Eastbourne, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Harrogate District Hospital, Harrogate, England
  - Kidderminster Hospital, Kidderminster Worcestershire, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Lincoln County Hospital, Lincoln, England
  - Cancer Research UK and University College London Cancer Trials Centre, London, England
  - Royal Marsden - London, London, England
  - St. Mary's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - King's Mills Hospital, Nottinghamshire, England
  - George Eliot Hospital, Nuneaton, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - Oldchurch Hospital, Romford, England
  - Conquest Hospital, Saint Leonards-on-Sea, England
  - Scarborough General Hospital, Scarborough, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Musgrove Park Hospital, Taunton, England
  - Torbay Hospital, Torquay, England
  - Warrington Hospital NHS Trust, Warrington, England
  - Warwick Hospital, Warwick, England
  - Sandwell General Hospital, West Bromwich, England
  - Weston General Hospital, Weston-super-Mare, England
  - West Cumberland Hospital, Whitehaven, England
  - New Cross Hospital, Wolverhampton, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil, England
  - Cancer Care Centre at York Hospital, York, England
  - Ninewells Hospital, Dundee, Scotland
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales